CLINICAL TRIAL: NCT00067236
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of Oral PG-116800 Following a Heart Attack
Brief Title: Study of Oral PG-116800 Following a Heart Attack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002135
Record Dates: First submitted 2003-08-13; First posted 2003-08-14 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-09

CONDITIONS: Myocardial Infarction; Heart Failure; Heart Enlargement
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Cardiomegaly | interventions — PG-116800

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PG-116800 tablet (Experimental): PG-116800 tablet (200 mg) taken twice daily for 90 days
  Interventions: Drug: PG-116800 (given as PG-530742)
- Placebo tablet (Placebo Comparator): Placebo tablet taken twice daily for 90 days
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: PG-116800 (given as PG-530742) — 200 mg tablet of PG-116800 (given as PG-530742)twice a day for 90 days
  Arms: PG-116800 tablet
Drug: Placebo tablet — placebo tablet, twice a day for 90 days
  Arms: Placebo tablet

SUMMARY:
The main purpose of the study is to test whether a possible new drug (called PG-116800) can prevent some of the damage to heart muscle in patients who have had a heart attack. The study will also supply information regarding possible uses of this compound in cardiovascular disease.

DETAILED DESCRIPTION:
Heart attacks cause damage to heart muscle that can weaken the heart and lead to changes in the shape and pumping ability of the heart. These changes can lead to heart failure. An enzyme called metalloproteinase (MMP) plays a role in this damage.

The main purpose of the study is to test whether a possible new drug (called PG-116800) that interferes with the MMP enzyme can prevent some of the damage to heart muscle in patients who have had a heart attack. The study will also supply information regarding possible uses of this compound in cardiovascular disease.

This is a Phase II "proof-of-concept" study; that is, it is a first attempt to treat sick people with the drug to see if it works.

The study is interventional since we will be using a drug to interfere with the heart tissue damage that follows a heart attack.

ELIGIBILITY:
Inclusion:

* Be at least 18 years of age but not older than 80 years of age at screening;
* Be diagnosed with a heart attack based on electrocardiogram (ECG) and cardiac enzymes criteria;
* The qualifying heart attack has to be a first heart attack;
* The qualifying heart attack has to result in a left ventricular ejection fraction (a measure of the working efficiency of the heart) between 15% and 40%.

Exclusion:

* Documented previous history of heart attack;
* Any past history of heart failure;
* Hemodynamic instability (no instability of circulatory system);
* History of congenital heart disease and cardiomyopathy (weakened heart muscle) associated with connective tissue disorders;
* Recent history or current moderate-to-severe kidney or liver impairment;
* Significant blood dyscrasias (disorders of the blood cells);
* Females who are currently: pregnant; breast-feeding; or are of childbearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2003-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Brum, MD, Study Director — Procter and Gamble
Locations (52):
- United States (21):
  - University of Arkansas for Medical Sciences and Central Arkansas Veterans Health Care System, Little Rock, Arkansas
  - Mercy Community Medical Center, Merced, California
  - Porter Adventist Hospital, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - JFK Medical Center, Atlantis, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Strong Memorial Hospital, Rochester, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Moses Cone Hospital, Greensboro, North Carolina
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Westmoreland Regional Hospital, Greensburg, Pennsylvania
  - Hershey Medical Center, Hershey, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Memorial Hermann Hospital, Houston, Texas
  - West Virginia University Hospital, Morgantown, West Virginia
- Canada (19):
  - Foothills Hospital, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Hospital, Edmonton, Alberta
  - Alder Medical Centre, Campbell River, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute, Victoria, British Columbia
  - St. John's HSC, Saint John's, New Brunswick
  - Queen Elizabeth II HSC, Halifax, Nova Scotia
  - Southlake Regional HC, Newmarket, Ontario
  - Scarborough Grace Hospital, Scarborough Village, Ontario
  - Toronto East General, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - CHUS, Hopital Fleurimont, Fleurimont, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Hopital Sacre-Coeur, Montreal, Quebec
  - Hopital Laval, Ste-Foy, Quebec
- Poland (12):
  - Klinika Kardiologii, Panstwowy Szpital Kliniczny, Bialystok, Bialystok
  - Katedra i Klinika Kardiologii i Chorob Wewnetznych, Akademia Medyczna w Bydgoszczy, Bydgoszcz, Bydgoszcz
  - 1 Katedra Kardiologii Slaskiej Akademii Medycznej, Katowice, Katowice
  - Klinika Chorob Serca i Naczyn, Krakowski Szpital Specjalistyczny, Krakow, Krakow
  - Oddzial Kardiologii, Wojewodzki Szpital Specjalistyczny, Krakow, Krakow
  - I Klinika Kardilogii Akademii Medycznej w Poznaniu, Poznan, Poznan
  - Oddzial Internistyczno-Kardiologiczny, Samodzieiny Publiczny Wojewodzki Szpital Zespolony, Szczecin, Szczecin
  - I Klinika Choroby Wiencowej, Instytut Kardiologii w Warszawie, Warsaw, Warszawa
  - Klinika Choroby Wiencowej, Instytut Kardiologi w Warszawie, Warsaw, Warszawa
  - Klinika Kardilogii Inwazyjnej, Centrainy Szpital MSWiA, Warsaw, Warszawa
  - Klinika Kardiologii, Szpital Grochowski, Warsaw, Warszawa
  - Klinika Kardiologii IMW, Uniwersytet Medyczny w Lodzi, Lodz, Łódź Voivodeship

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet twice daily for 90 days
- PG-116800 Tablet: PG-116800 tablet (200 mg) twice daily for 90 days
Period: Overall Study
Arm/Group | Placebo | PG-116800 Tablet
Started | 128 | 125
Completed | 108 | 99
Not Completed | 20 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PG-116800 Tablet | Total
Number analyzed (Participants) | 128 | 125 | 253
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (10.22) | 59.7 (11.71) | 59.8 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 94 | 93 | 187
Region of Enrollment [Number; unit: participants]
  United States | 19 | 16 | 35
  Canada | 22 | 23 | 45
  Poland | 87 | 86 | 173

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVi in mL/m2) at Day 90 Post Myocardial Infarction (MI)
Description: Mean change of left ventricular end diastolic volume index (mL/m2) as evaluated via ventricular end-diastolic volume index augmentation 90 days post Myocardial Infarction (MI)
Time Frame: 90 days
Population: A patient was considered evaluable for the primary efficacy assessment if data were complete for at least the baseline and Day 90 visit (i.e., no data were imputed for the primary endpoint).
Measure: Mean (Standard Error); unit: mL/m2
Arm/Group | Placebo | PG-116800 Tablet
Number analyzed (Participants) | 108 | 99
mL/m2 | 5.48 (1.41) | 5.09 (1.45)
Statistical Analysis 1: Comparison: Placebo vs PG-116800 Tablet; Changes from baseline in efficacy parameters at Day 90; Test type: Superiority or Other; p = 0.4239, ANOVA; Mean Difference (Net) = 4

ADVERSE EVENTS:
Arm/Group | Placebo | PG-116800 Tablet
Serious Adverse Events (participants affected / at risk) | 67/128 | 75/125
Other Adverse Events (participants affected / at risk) | 124/128 | 124/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | PG-116800 Tablet (N=125)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure NOS (Cardiac disorders) | 7 (9) | 3 (5)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 6 (8)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 3 (3)
Acute coronary sydrome (Cardiac disorders) | 3 (3) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 7 (7)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vestibular neruontis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
oedema peripheral (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 3 (3) | 2 (2)
Discomfort (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions (General disorders) | 5 (5) | 4 (4)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis acute (Infections and infestations) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedemas (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Face oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis medicamentosa (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular pesuoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | PG-116800 Tablet (N=125)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (5)
Fatigue (General disorders) | 9 (10) | 0 (0)
Pyrexia (General disorders) | 9 (10) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 17 (29)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 4 (6) | 6 (7)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (12) | 7 (10)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Headache (Nervous system disorders) | 11 (11) | 7 (9)
Dizziness (Nervous system disorders) | 11 (11) | 3 (5)
Anxiety (Nervous system disorders) | 2 (2) | 8 (8)
Insomnia (Nervous system disorders) | 12 (13) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 10 (10)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 13 (13)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Hypertension (Vascular disorders) | 10 (14) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data, calculations, interpretations, opinions, and recommendations will be the property of P&GP. Manuscripts for publication will be drafted by the Expert Panel which will select appropriate journals in which to publish. P&GP, through its Expert Panel representation, will provide technical/editorial/review assistance. Other manuscript(s) will supported as appropriate. These materials must be submitted to P&GP and the Expert Panel for review prior to publication